CLINICAL TRIAL: NCT02711761
Title: Ideal Depth of Guide Wire for Right Internal Jugular Vein During Central Line Insertion
Brief Title: Ideal Depth of Guide Wire for Central Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-2015-105
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Patient Safety During Central Venous Catheterization
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- 15 cm (Experimental): The depth of guide wire will be 15 cm from puncture site of skin prior to tissue dilation during central venous catheterization
  Interventions: Device: central venous catheterization
- 17.5 cm (Experimental): The depth of guide wire will be 17.5 cm from puncture site of skin prior to tissue dilation during central venous catheterization
  Interventions: Device: central venous catheterization
- 20 cm (Active Comparator): The depth of guide wire will be 20 cm from puncture site of skin prior to tissue dilation during central venous catheterization
  Interventions: Device: central venous catheterization

INTERVENTIONS:
Device: central venous catheterization — 15 cm: The depth of guide wire prior to tissue dilation during central venous catheterization will be 15 cm.
  17.5 cm: The depth of guide wire prior to tissue dilation during central venous catheterization will be 17.5 cm.
  20 cm: The depth of guide wire prior to tissue dilation during central venous catheterization will be 20 cm.

SUMMARY:
prospective randomized double-blind controlled study

DETAILED DESCRIPTION:
Total of 69 ASA (American Society of Anesthesiologist) physical status class I or II patients will be enrolled.

Randomly assigned to three group according to the depth of guide-wire prior to tissue dilation during central catheterization via right internal jugular vein. (Group 1: 15 cm / Group 2: 17.5 cm / Group 3: 20 cm)

Central catheterization will be performed by anesthesiologists who be blinded to this study protocol.

An investigator will monitor and record whether any arrhythmia will occur.

The incidence of occurrence of arrhythmia will be compared between three groups.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving general anesthesia requiring central venous catheterization via right internal jugular vein.
* ASA (American Society of Anesthesiologist) physical status class I or II

Exclusion Criteria:

* at the pre-anesthetic evaluation, history of any arrhythmia
* when monitoring before the induction of anesthesia in the operating room, newly arrhythmia is observed.
* abnormal electrolyte at the pre-anesthetic evaluation
* too difficult to access right internal jugular vein for central catheterization (too short neck, infection at the site of right internal jugular vein, ventriculoperitoneal shunt or chemo-port existence at the site of right internal jugular vein. too close site to operating field)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of arrhythmia | during central venous catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D., Study Director — Seoul National University Boramae Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, Seoul, South Korea